CLINICAL TRIAL: NCT06069830
Title: PET and EBV DNA-directed Therapy for Localized Nasal Extranodal NK/T Cell Lymphoma
Acronym: ENKTL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PENK
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: NK-T-Cell Lymphoma, Extranodal
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interim PET and EBV DNA-directed therapy (Experimental): According to the interim PET and EBV DNA results, patients are divided into three cohorts: 1) cohort A: Deauville score 1-3 and EBV DNA negativity; 2) cohort B: Deauville score 1-3 and EBV DNA positivity; 3) cohort C: Deauville score 4-5.
  Interventions: Drug: 4 cycles of ESA regimen with sandwiched radiotherapy; Drug: 2 cycles of ESA regimen sequential radiotherapy and 2 cycles of PD-1 monoclonal antibody combined with pegaspargase; Drug: 2 cycles of ESA regimen, 2 cycles of PD-1 monoclonal antibody and concurrent radiotherapy, 2 cycles of PD-1 monoclonal antibody combined with pegaspargase

INTERVENTIONS:
Drug: 4 cycles of ESA regimen with sandwiched radiotherapy — Pegaspargase, 2500U/m2, i.m. d1; etoposide, 200mg, p.o., d2-d4; Dexamethasone, 40mg, p.o. d2-d4；
Drug: 2 cycles of ESA regimen sequential radiotherapy and 2 cycles of PD-1 monoclonal antibody combined with pegaspargase — Pegaspargase, 2500U/m2, IM, d1; PD-1 monoclonal antibody, 200mg, i.v. d2;
Drug: 2 cycles of ESA regimen, 2 cycles of PD-1 monoclonal antibody and concurrent radiotherapy, 2 cycles of PD-1 monoclonal antibody combined with pegaspargase — PD-1 monoclonal antibody, 200mg, i.v. d1

SUMMARY:
A prospective, open-abel, phase 2 clinical study to investigate whether interim Positron Emission Tomography (PET) and Epstein-Barr virus (EBV) DNA-directed therapy can improve the prognosis of localized nasal extranodal NK/T cell lymphoma (ENKTL) patients.

DETAILED DESCRIPTION:
This study aims to evaluate the significance of mid-term PET and EBV DNA-directed therapy for localized nasal ENKTL. Patients receive 2 cycles of ESA (Pegaspargase, Etoposide, Dexamethasone) regimen, then according to the mid-term PET and EBV DNA results, patients are divided into three cohorts: 1) cohort A: patients with Deauville score 1-3 and EBV DNA negative receive sequential radiotherapy and 2 cycles of ESA regimen; 2) cohort B: patients with Deauville score 1-3 and EBV DNA positive receive sequential radiotherapy and 2 cycles of PD-1 monoclonal antibody combined with pegaspargase; 3) cohort C: patients with Deauville score 4-5 receive 2 cycles of PD-1 monoclonal antibody and concurrent radiotherapy, then 2 cycles of PD-1 monoclonal antibody combined with pegaspargase.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically newly diagnosed extranodal NK/T cell lymphoma, nasal type (according to the WHO classification 2016);
* No previous anti-lymphoma treatment;
* Age ≥ 18 years old;
* Ann Arbor stage I/II;
* ECOG 0-2 score;
* Patients with a life expectancy of at least 3 months;
* At least one measurable / evaluable lesion from diagnostic biopsy to the beginning of treatment;
* Sufficient bone marrow and liver and kidney function, namely:

  1. Absolute neutrophil count (ANC)> 1000 / μL, platelet count> 50, 000 / μl, hemoglobin> 9g/ dl;
  2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <3 times the upper limit of normal (ULN); Serum total bilirubin <1. 5 times ULN (patients with Gilbert syndrome can be included);
  3. Serum creatinine <2 times ULN or creatinine clearance rate> 50 ml/min.
* Able to comply with the research procedures and cooperate in the implementation of the entire research process;
* Written informed consent;
* Women with fertility agree to take appropriate measures to avoid pregnancy during the treatment period until at least one year after the end of treatment; Men agree to maintain abstinence or use barrier contraception.

Exclusion Criteria:

* Diagnosed invasive NK cell leukemia and extranasal ENKTL;
* Ann Arbor stage III/IV;
* Pregnant or lactation;
* Autoimmune diseases that require systemic treatment in the past 2 years (namely, antirheumatic drugs, hormones or immunosuppressants), including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome related vascular thrombosis, Wegener's granuloma, Sjogren's syndrome, Guillain Barre syndrome, multiple sclerosis, vasculitis or glomerulonephritis. The following cases are allowed to be included: autoimmune hypothyroidism or type I diabetes receiving stable treatment, hormone replacement treatment (such as thyroxine, insulin, or supplement of physiological hormone due to insufficient adrenal or pituitary gland) are not considered as systematic treatment and are allowed to be included.
* Other invasive cancers that have not received curative treatment or are still receiving anti-cancer treatment (including hormone therapy for breast cancer or prostate cancer) in the past 3 years;
* Pneumonia requiring steroid medication treatment (non-infectious); Or had clinical evidence of interstitial lung disease or active and non-infectious pneumonia;
* Active infections that require systemic treatment;
* Severe cardiovascular disease, or myocardial infarction, unstable arrhythmia, or unstable angina pectoris occurring 3 months ago;
* Previous treatment with anti PD-1, anti PD-L1, or anti PD-L2 drugs;
* HBsAg, HCV, or HIV positivity; HBV and HCV serological positivity is allowed, but DNA/RNA must be negative;
* Live attenuated vaccine vaccination within 4 weeks before the treatment; patients are prohibited from receiving live attenuated vaccines during the study period, including influenza vaccines;
* Central nervous system diseases;
* Previous allogeneic tissue/solid organ transplantation;
* Active tuberculosis;
* Other concurrent uncontrollable medical conditions that may interfere the participation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival rate | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
2-year overall survival rate | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.
2-year PFS and OS rates in the subgroups of interim Deauville score 1-3 with EBV DNA negative, Deauville 1-3 with EBV DNA positive, and Deauville 4-5 | Baseline up to data cut-off (up to approximately 2 years)
  PFS was progression-free survival; OS was overall survival.
Objective response rate | End of treatment (6-8 weeks after last cycle)
  Percentage of participants with complete response and partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Complete response rate | End of treatment (6-8 weeks after last cycle)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Treatment-Related Adverse Events rate as assessed by CTCAE version 5.0 | From enrollment to study completion, a maximum of 3 years
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Changes of plasma EBV DNA load | From enrollment to study completion, a maximum of 3 years
  Plasma EBV DNA load monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China